CLINICAL TRIAL: NCT05692011
Title: The Effects of a AN69ST Membrane and Polysulphone Membrane on Septic Children With Continuous Blood Purification
Brief Title: AN69ST Verse PS in CBP in Septic Children
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: West China Second University Hospital (Other); Children's Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Shandong Provincial Hospital (Other Government); Children's Hospital of Soochow University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-28
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sepsis
Keywords: sepsis; blood purification
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the volume of 2ml whole blood was stored in EDTA tube
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- blood purification(AN69ST)
  Interventions: Device: blood purification(AN69ST)
- blood purification(PS)
  Interventions: Device: blood purification(PS)

INTERVENTIONS:
Device: blood purification(PS) — After the sepsis patients were enrolled, they were treated with blood purification in CVVH mode with PS membrane, 24 hours per day, for 3 consecutive days
  Groups: blood purification(PS)
Device: blood purification(AN69ST) — After the sepsis patients were enrolled, they were treated with blood purification in CVVH mode with AN69ST membrane, 24 hours per day, for 3 consecutive days
  Groups: blood purification(AN69ST)

SUMMARY:
In septic shock, dysregulated host responses to pathogens lead to cytokine storms that damage host tissues and organs, further contributing to the development of organ dysfunction and increased mortality. For sepsis, blood purification can remove inflammatory factors in sepsis by filtration or adsorption, so as to achieve the purpose of reducing inflammatory mediators in the body. However, there are few prospective randomized controlled studies in children. Therefore, this study intends to compare the efficacy and prognosis of different membrane on children with sepsis through a perspective cohort study, so as to provide a corresponding basis for the treatment of children with sepsis blood purification.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction resulting from a dysregulated host response to infection. In septic shock, dysregulated host responses to pathogens lead to cytokine storms that damage host tissues and organs, further contributing to the development of organ dysfunction and increased mortality.

Blood purification therapy is gradually developed on the basis of renal replacement therapy, and now it is more and more widely used in the field of critical care in children. CVVH can reduce the level of inflammation in the body in different membranes, but the results of reducing inflammatory factors are different, and the outcomes of patients are also different.

Blood purification treatment can reduce inflammatory mediators in sepsis, but there are few prospective randomized controlled studies in children. Therefore, this study intends to compare the efficacy and prognosis of different blood purification membrane in children with sepsis through a perspective cohort study. Provide the corresponding basis for blood purification treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2005 diagnostic criteria for sepsis
* Age 29 days - 18 years old
* Sepsis-induced dysfunction of more than one organ or abnormal tissue perfusion, or septic shock
* Diagnosis < 48 hours

Exclusion Criteria:

* Inability to obtain an informed consent from the subject, family member or an authorized surrogate
* Subject has end-stage renal disease and requires chronic dialysis
* There is clinical support for non-septic shock
* Subject has had chest compressions as part of cardiopulmonary resuscitation this hospitalization without immediate return to communicative state
* Subject has uncontrolled hemorrhage
* Subject has immunodeficiency diseases
* Subject has received chemoradiotherapy or immunosuppressive therapy in the 14 days before enrollment
* HIV infection in association with a last known or suspected CD4 count of <50/mm3
* Subject has sustained extensive third-degree burns within the past 7 days
* Subject has known sensitivity or allergy to heparin or has a history of heparin associated thrombocytopenia
* Subject is currently enrolled in an investigational drug or device trial
* Subject has been previously enrolled in the current trial
* Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment, such as end stage chronic illness with no reasonable expectation of survival to hospital discharge
* Known hypersensitivity to hemofilter
* Subject has received organ transplantation
* Subject is expected to die within 24 hours

Ages: 29 Days to 28 Years | Sex: All
Age Groups: Child, Adult
Study Population: children with sepsis requiring blood purification
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cytokine change | from enrollment to the 3th days
  This is a binary variable. It is also a compositional variable including IL-6, IL-10, TNF-a, IL-4, IL-2 and etc. If one of the factors changes, it is considered that the variable changes. If the cytokine drops below half of the original value, it is considered to be changed. The cytokine would be measured measured at the 7th day after enrollment
organ injury changes | from enrollment to the 3th days
  the difference of the organ injury changes would be measured at the 3th day after enrollment

SECONDARY OUTCOMES:
survival rate | from enrollment to the 28th days
  the survival rate would be measured at the 28th day after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Of Soochow University, Suzhou, China